CLINICAL TRIAL: NCT03051191
Title: Exploring the Pathogenic Mechanisms Shared by Cancer and Cardiovasuclar Diseases
Brief Title: Pathogenic Mechanisms of Cancer and Cardiovascular Diseases
Status: Completed | Type: Observational
Sponsor: Sakakibara Heart Institute (Other)
Collaborators: Japanese Foundation for Cancer Research (Other)
Responsible Party: Sponsor
Other Study IDs: SHIP02
Record Dates: First submitted 2017-02-09; First posted 2017-02-13 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2017-02

CONDITIONS: Pathogenesis; Cardiovascular Diseases; Cancer
Keywords: atherosclerotic cardiovascular diseases; nonischemic heart failure; cancer
MeSH Terms: conditions — Cardiovascular Diseases; Neoplasms | interventions — Noninvasive Prenatal Testing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — plasma containing cell free DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- 1: No ACVD/NIHF or cancers: The patients who do not have ACVD, NIHF or cancers
  Interventions: Diagnostic Test: micro RNA
- 2: Cancers but no ACVD/NIHF: The patients who have cancers but no ACVD/NIHF
  Interventions: Diagnostic Test: micro RNA
- 3: ACVD and cancers: The patients who have ACVD and cancers
  Interventions: Diagnostic Test: micro RNA
- 4: ACVD but no cancers: The patients who have ACVD but no cancers
  Interventions: Diagnostic Test: micro RNA
- 5: NIHF and cancers: The patients who have NIHF and cancers
  Interventions: Diagnostic Test: micro RNA
- 6: NIHF but no cancers: The patients who have NIHF but no cancers
  Interventions: Diagnostic Test: micro RNA

INTERVENTIONS:
Diagnostic Test: micro RNA — micro RNA, cell free DNA and 16S rRNA genes will be explored cross-sectionally at enrollment.
  Other Names: cell free DNA; 16S rRNA genes of gut microbiota

SUMMARY:
Subjects with cardiovascular diseases (CVD) have higher incidence of cancers compared to general population. The investigators hypothesized that shared molecular mechanism play a pivotal role in the pathogenesis of CVD including heart failure (HF) and cancers. To address this hypothesis, the investigators are going to explore the expression pattern of micro RNA (miRNA) and cell free DNA (cfDNA) derived from host, gut microbiota and gut microbiota composition extensively in patients with or without CVD, non-ischemic HF (NIHF), and cancers. The participants will be recruited from the outpatient clinic in Sakakibara Heart Institute or Japanese Foundation for Cancer Research. By comparing the expression pattern of miRNA, cfDNA, or gut microbiota composition, the investigators are seeking to find the pathogenic mechanisms shared by those diseases.

DETAILED DESCRIPTION:
It has been reported that subjects with cardiovascular diseases (CVD) have higher incidence of cancers compared with general population. Because of the genetic and traditional commonalities between the underlying causes of CVD and cancers, the investigators hypothesized that shared molecular mechanism play a pivotal role in the pathogenesis of CVD including heart failure (HF) and cancers.

MicroRNAs (miRNAs) are small, single-stranded non-coding RNA sequences of about 18-22 nucleotides that interact with specific target messenger RNAs. They are known to be involved in the various processes including development, homeostasis, cell differentiation, proliferation, apoptosis and various diseases by modulating post-transcriptional and translational processes. Some of miRNAs have been reported to be involved in the pathogenesis of cancers. Cell free DNAs (cfDNA) is extracellular nucleic acids found in cell-free plasma in humans. Elevated level of cfDNA was reported in patients with cancer and CVD. 16S ribosomal RNA (rRNA) genes are distinct in microbiota, which can be utilized to quantify the bacterial DNA in the systemic circulation. 16S rRNA genes are also shown to be elevated in patients with CVD. These findings imply the possibility that translocated microbiota might play pivotal roles in the pathogenesis of CVD and cancers. The quantity and composition of gut microbiota have been shown to be altered in various diseases including obesity, diabetes mellitus, hypertension and CVD. The previous findings from fecal transplantation experiments, which showed the disease phenotype was transferred from one to another subject (animal or human), strongly suggest the possibility that microbiota play some pathogenic roles in those diseases.

To address this hypothesis, the investigators are going to cross-sectionally explore the expression pattern of miRNA and cfDNA and the composition of gut microbiota extensively in patients with or without atherosclerotic CVD (ACVD), non-ischemic HF (NIHF), and cancers. The investigators will recruit the participants from the patients who regularly visit the outpatient clinic in Sakakibara Heart Institute or The Cancer Institute Hospital of Japanese Foundation of Cancer Research. The investigators will recruit the patients without ACVD or NIHF and with/without cancers (Group 1/2), those with ACVD and with/without cancers (Group 3/4), and those with NIHF and with/without cancers (Group 5/6). Their peripheral blood will be drawn and stools will be collected. miRNA in exosome will be extracted from plasma and explored by miRNA microarray. cfDNA pattern will be extensively explored by microarray. By comparing the expression pattern of miRNA and cfDNA, and the composition of gut microbiota by 16s rRNA gene shotgun analysis, the investigators will be seeking to find the molecular mechanisms shared by those diseases.

ELIGIBILITY:
Inclusion Criteria:

* subjects who regularly visit outpatient clinic in Sakakibara Heart Institute or The Cancer Institute Hospital of Japanese Foundation of Cancer Research.

Exclusion Criteria:

* subjects who have multiple cancers

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who regularly visit outpatient clinic in Sakakibara Heart Institute or The Cancer Institute Hospital of Japanese Foundation of Cancer Research.
Sampling Method: Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
miRNA | At enrollment
  Expression pattern of miRNA in blood
Cell free DNA from host | At enrollment
  Quantity of cell free DNA derived from host in blood
Cell free DNA from microbiota | At enrollment
  Expression pattern of cell free DNA distinct from microbiota in blood
bacterial composition in stool | At enrollment
  the bacterial composition analyzed by shot gun analysis of 16s rRNA genes in stool

CONTACTS AND LOCATIONS:
Overall Officials: Tsutomu Yoshikawa, Principal Investigator — Sakakibara Heart Institute
Locations (2):
- Japan (2):
  - Sakakibara Heart Institute, Fuchū
  - The Cancer Institute Hospital for Japanese Foundation for Cancer Research, Tokyo

IPD SHARING:
Plan to Share IPD: No